CLINICAL TRIAL: NCT01612117
Title: Is Urinary Neutrophil Gelatinase-Associated Lipocalin (uNGAL) the "Renal Troponin" in Invasive Cardiology?
Brief Title: Urinary Neutrophil Gelatinase-Associated Lipocalin (uNGAL) in Invasive Cardiology
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Stéphane Cook, Prof, Ms, University of Freiburg
Other Study IDs: 013-REP-CER-FR
Record Dates: First submitted 2012-05-30; First posted 2012-06-05 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Renal Failure
Keywords: renal failure; cardiology; contrast-induced nephropathy
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urinary samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- consecutive, PCP patients: All patients requiring percutaneous coronary procedures, such as coronary angiography or intervention

SUMMARY:
Diagnosis of acute kidney injury (AKI) relies on a late marker, namely serum creatinine (SCr). New biomarkers are considered for early and sensitive detection of CIN. In particular, uNGAL has been used for early detection of AKI in the emergency department, after cardiopulmonary bypass or following CM administration.

This study will be conducted to assess the possible value of urinary Neutrophil Gelatinase-Associated Lipocalin (uNGAL) as an early detector of contrast-induced nephropathy (CIN) in a large sized cohort of patients undergoing percutaneous coronary procedures (PCP) and whether or not uNGAL correlates with the volume of contrast medium (CM) used.

DETAILED DESCRIPTION:
Methods. We will enroll all consecutive patients undergoing PCP with iomeprolum during a 3-month period at our institution. CIN will be defined as a ≥25% increase in SCr from baseline when measured 2-4 days after PCP. uNGAL will be measured at its peak with the Abbott ARCHITECT assay.

ELIGIBILITY:
Inclusion Criteria:

* All except patients with exclusion criteria

Exclusion Criteria:

* dialysis-dependent chronic kidney disease
* lack of written consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
to assess the value of uNGAL measurement 4 to 6 hours after PCP as a possible early detector of CIN | 4-6 hours after PCP
  cf title

SECONDARY OUTCOMES:
to study the relationship between the volume of contrast medium used for PCP and the uNGAL levels measured 4 to 6 hours thereafter | 4-6 hours after PCP
  cf. title

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Cook, MD, Study Chair — University Fribourg
Locations (1):
- Department of Cardiology, Fribourg, Canton of Fribourg, Switzerland

REFERENCES:
- [Result] Perrin T, Descombes E, Magnin JL, Gachet M, Hemett OM, Hayoz D, Stolt V, Baeriswyl G, Stauffer JC, Goy JJ, Togni M, Cook S. Urinary Neutrophil Gelatinase-Associated Lipocalin (uNGAL) and contrast-induced acute kidney injury after coronary angiogram. Swiss Med Wkly. 2013 Aug 27;143:w13853. doi: 10.4414/smw.2013.13853. eCollection 2013. PMID 23986375